CLINICAL TRIAL: NCT03007394
Title: Phase 2, Multi-Center Trial of Lorcaserin in the Treatment of Cocaine Use Disorder
Brief Title: Lorcaserin in the Treatment of Cocaine Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA/VACSP #1033
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-02

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Use Disorder
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorcaserin (Active Comparator): 10 mg capsule by mouth, twice a day, for 13 weeks
  Interventions: Drug: Lorcaserin
- Placebo Oral Capsule (Placebo Comparator): 10 mg placebo capsule, twice a day, for 13 weeks
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin Capsule
  Other Names: Belviq; lorcaserin hydrochloride
  Arms: Lorcaserin
Drug: Placebo Oral Capsule — sugar pill to mimic lorcaserin 10mg capsule
  Arms: Placebo Oral Capsule

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of lorcaserin in the treatment of cocaine use disorder.

DETAILED DESCRIPTION:
This is a 19-week, multi-center, randomized, Phase 2 clinical study comparing the efficacy of lorcaserin (10mg, b.i.d) to matched placebo in the treatment of cocaine use disorder. Up to 3 weeks will be allowed for the Screening Period and a 13-week treatment phase, with a 3-week follow-up period, with scheduled visits during Study weeks 14 and 16.

ELIGIBILITY:
Inclusion Criteria:

* Has a DSM-5 diagnosis of current cocaine use disorder as verified by the Structured Clinical Interview for DSM-5
* Is seeking treatment for cocaine use disorder
* Is able to understand and provide written informed consent
* Has used cocaine on at least 1 day in the last 30 days prior to screening
* Has completed all psychological assessments and procedures during the screening period
* If female, not pregnant, lactating, unable to conceive OR must agree to use an acceptable method of birth control
* Has a total body weight greater than 110 pounds and body mass index greater than 20

Exclusion Criteria:

* Contact site for more information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shwe Gyaw, MD, Study Chair — National Institute on Drug Abuse (NIDA)
Locations (12):
- United States (12):
  - Pacific Treatment and Research Center, La Jolla, California
  - Matrix Institute on Addictions, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - George Washington University, Washington D.C., District of Columbia
  - Meridien Research, Lakeland, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Boston University School of Medicine, Boston, Massachusetts
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Neuro-Behavioral Clinical Research Inc., Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - CODA, Inc., Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lorcaserin | Placebo Oral Capsule
Started | 118 | 154
Completed | 91 | 91
Not Completed | 27 | 63

BASELINE CHARACTERISTICS:
Population: The "Intent-to-Treat (ITT) Population" of 272 are all subjects who may have taken at least one dose of lorcaserin or placebo after randomization.
  2) The "PPEE Population" of 242 is the subset of the ITT Population who pre-qualify for the primary efficacy endpoint by meeting the specified PPEE criteria prior to randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin | Placebo Oral Capsule | Total
Number analyzed (Participants) | 118 | 124 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.88) | 50.3 (9.99) | 50.2 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 40 | 68
  Male | 90 | 84 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 109 | 113 | 222
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 77 | 83 | 160
  White | 35 | 30 | 65
  More than one race | 4 | 9 | 13
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 118 | 124 | 242

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Actual Number of Subjects That Successfully Achieve Abstinence From Cocaine During the Last Three Weeks of Treatment in the "Pre-qualified for Primary Efficacy Endpoint" (PPEE) Population
Description: Self-report data indicating no cocaine use on each day of the 3-week period, at least one benzoylecgonine (BE) assay result for a urine sample collect within the 3-weeks period and BE assay results are negative for all urine samples collected during the 3-week period.
Time Frame: Treatment weeks 11 - 13
Measure: Number; unit: participants
Arm/Group | Lorcaserin | Placebo Oral Capsule
Number analyzed (Participants) | 118 | 124
participants | 1 | 4

2. Secondary Outcome: The Secondary Endpoint is the Actual Number of Subjects That Successfully Achieve Abstinence From Cocaine During the Last Three Weeks of Treatment Who Are Either Non-Drinkers or Who Are Attempting Alcohol Abstinence
Time Frame: Treatment weeks 11-13
Measure: Number; unit: participants
Arm/Group | Lorcaserin | Placebo Oral Capsule
Number analyzed (Participants) | 118 | 124
participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every week during treatment and through study follow-up, a 13-week treatment phase with a 4-week follow-up period.
Description: 1. The "Intent-to-Treat (ITT) Population" of 272 are all subjects who may have taken at least one dose of lorcaserin or placebo after randomization as noted in the total for the participant flow.
  2. The "PPEE Population" of 242 is the subset of the ITT Population who pre-qualify for the primary efficacy endpoint by meeting the specified PPEE criteria prior to randomization, which is the subset population used here
Arm/Group | Lorcaserin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/124
Serious Adverse Events (participants affected / at risk) | 4/118 | 6/124
Other Adverse Events (participants affected / at risk) | 66/118 | 69/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin (N=118) | Placebo Oral Capsule (N=124)
Hospitalization (General disorders) | 2 | 6
Life threatening and hospitalization (Cardiac disorders) | 1 | 0
Life threatening and hospitalization (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin (N=118) | Placebo Oral Capsule (N=124)
Blood pressure increase/decrease (Investigations) | 14 | 19
Abdominal Distress (Gastrointestinal disorders) | 20 | 18
Infection (Infections and infestations) | 16 | 21
Headache (Nervous system disorders) | 19 | 13
Body pain (Musculoskeletal and connective tissue disorders) | 8 | 18
Depression/Anxiety (Psychiatric disorders) | 16 | 11
Fatigue (General disorders) | 13 | 13
Rash (Skin and subcutaneous tissue disorders) | 11 | 7
Bodily injury (Injury, poisoning and procedural complications) | 8 | 8
Hypertension (Vascular disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT03007394/Prot_SAP_000.pdf